CLINICAL TRIAL: NCT01778270
Title: Not Invasive Monitoring of Pleural Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-078
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; pleural drainage; thorax impedance; respiration parameters; heart sounds analysis
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non invasive sensor pleural drainage (Other): feasibility data will be collected with thorax impedance measurements via body bioimpedance sensor in Ohm before and after pleura drainage, via impedance cardiography stroke volume and cardiac output will be calculated and also respiratory parameters determined via capnograph as carbon dioxide (CO2) in %/ml exhaled volume before and after pleura drainage. Additionally heart sound analysis via electronic stethoscope will be compared to standard methods.
  Interventions: Device: Body Bioimpedance Sensor
- non invasive sensor healthy control (Other): the same measurements as in arm 1: feasibility data will be collected with thorax impedance measurements via body bioimpedance sensor before and after pleura drainage in Ohm, via impedance cardiography stroke volume and cardiac output will be calculated and also respiratory parameters determined via capnograph as carbon dioxide (CO2) in %/ml exhaled volume once in 25 healthy controls.
  Additionally heart sound analysis via electronic stethoscope will be compared to standard methods.
  Interventions: Device: Body Bioimpedance Sensor

INTERVENTIONS:
Device: Body Bioimpedance Sensor

SUMMARY:
This study investigates if data about monitoring the drainage of pleural effusion can be collected by non invasive sensors (feasibility).

DETAILED DESCRIPTION:
25 patients > 18 years old with pleura effusion will be examined with regard to the feasibility of non invasive sensor measurements corresponding to the course of thorax impedance and respiration parameters during body fluids loss before and after pleural drainage. The measured data will be compared to standard routine reference measurements (heart rate, medication, brain natriuretic peptide (BNP), heart minute volume). Additionally heart sound analysis via electronic stethoscope will be compared to standard methods.

Also 25 healthy controls will undergo the same measurements to receive standard values.

ELIGIBILITY:
Inclusion Criteria:

* patients with pleural effusion undergoing pleural drainage
* male and female patients aged at least 18 years

Exclusion Criteria:

* pregnancy or breast feeding
* implanted pacemaker / Cardiac Resynchronization Therapy (CRT) / Implanted Cardioverter Defibrillator (ICD) except Medtronic Device "OptiVol".
* patients not being able to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change of thorax impedance (Ohm) | once during hospital stay at baseline time 0 before pleura drainage and after pleura drainage at time 1 hour.
  non invasive bioimpedance measurements to determine feasibility of body fluid loss before and after pleura drainage in 25 patients > 18 years old; also 25 healthy controls are measured to receive standard values

SECONDARY OUTCOMES:
Change of Cardiac output ( l/min) via impedance cardiography | once during hospital stay at baseline time 0 before pleura drainage and after pleura drainage at time 1 hour
  non invasive bioimpedance measurements to determine feasibility of impedance cardiography before and after pleura drainage; also 25 healthy controls are measured to receive standard values

OTHER OUTCOMES:
Change of respiratory parameter CO2 in %/ml exhaled air | once during hospital stay at baseline time 0 before pleura drainage and after pleura drainage at time 1 hour
  respiratory parameters as CO2 in %/ml exhaled volume will be determined via capnograph

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Marx, MD, Study Director — Medical Clinic I, University Hospital Aachen
Locations (1):
- Univeristy Hospital Aachen, Aachen, North Rhine Westfalia, Germany

REFERENCES:
- [Derived] Zink MD, Weyer S, Pauly K, Napp A, Dreher M, Leonhardt S, Marx N, Schauerte P, Mischke K. Feasibility of bioelectrical impedance spectroscopy measurement before and after thoracentesis. Biomed Res Int. 2015;2015:810797. doi: 10.1155/2015/810797. Epub 2015 Mar 11. PMID 25861647